CLINICAL TRIAL: NCT01945385
Title: Impact of Video Intervention on Postabortal Uptake of Long Acting Reversible Contraception (LARC)
Acronym: LARC IUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 13-0185
Record Dates: First submitted 2013-07-29; First posted 2013-09-18 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Abortion
Keywords: Abortion; LARC; Contraception; IUD; Contraceptive implant; behavioral change; video intervention

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video intervention (Experimental): Participants will view a seven - minute theory-based video of patient testimonials about their own postabortal LARC uptake.
  Interventions: Behavioral: Video intervention
- Control (No Intervention): Patients will view a 7 minute video about stress management delivered by local psychologist.

INTERVENTIONS:
Behavioral: Video intervention — Brief 7 minute video of physician describing LARC methods followed by two patient testimonials about their own postabortal LARC experience.
  Arms: Video intervention

SUMMARY:
Primary: To compare rates of immediate postabortal LARC uptake between women exposed to a brief, theory-based, video intervention prior to standard contraceptive counseling and women exposed to standard counseling alone.

Secondary: To identify predictors of immediate postabortal LARC uptake among all participants including the role of:

* Demographic and reproductive health history variables
* Baseline decisional balance, self-efficacy and stage of change for contraceptive initiation

DETAILED DESCRIPTION:
This is a randomized controlled trial evaluating the effect of a brief video intervention on postabortal uptake of long acting reversible contraception.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 29 Surgical abortion being performed the day of the study English speaking

Exclusion Criteria:

* Nonviable pregnancy Sexual assault Administered sedative medication Non English speaking

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 193 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Postabortal LARC uptake | Immediate
  Immediate uptake of IUD or contraceptive implant following surgical abortion

SECONDARY OUTCOMES:
Perceived self efficacy surrounding LARC decision making | Baseline
  Subject's own perception of her ability to uptake LARC in the postabortal period.
Perceived decisional balance surrounding LARC decision making | Immediate
  Subjects perceived pros and cons around starting a LARC method in the postabortal period
Stage of behavioral change around LARC uptake | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Gilliam, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- Planned Parenthood Near North, Chicago, Illinois, United States